CLINICAL TRIAL: NCT01732510
Title: A Phase Ib Randomized, Double-Blinded, Placebo-Controlled Multiple Rising Dose Clinical Trial to Evaluate the Safety, Efficacy, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Intravenous MK-8226 in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Intravenous MK-8226 in Participants With Moderate-to-Severe Atopic Dermatitis (MK-8226-003)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was prematurely stopped due to business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8226-003; 2012-005560-95 (EudraCT Number)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1: MK-8226 0.3 mg/kg (Experimental): MK-8226 administered intravenously (IV) at a weight-based dose every 2 weeks for a period of 12 weeks.
  Interventions: Drug: MK-8226
- Part 1: MK-8226 1 mg/kg (Experimental): MK-8226 administered IV at a weight-based dose every 2 weeks for a period of 12 weeks.
  Interventions: Drug: MK-8226
- Part 1: MK-8226 3 mg/kg (Experimental): MK-8226 administered IV at a weight-based dose every 2 weeks for a period of 12 weeks.
  Interventions: Drug: MK-8226
- Part 1: MK-8226 10 mg/kg (Experimental): MK-8226 administered IV at a weight-based dose every 2 weeks for a period of 12 weeks.
  Interventions: Drug: MK-8226
- Part 1: Placebo (pooled) (Placebo Comparator): Dose-matched placebo administered IV every 2 weeks for a period of 12 weeks.
  Interventions: Drug: Placebo
- Part 2: MK-8226 3 mg/kg (Experimental): MK-8226 administered IV at a weight-based dose every 2 weeks for a period of 12 weeks.
  Interventions: Drug: MK-8226
- Part 2: Placebo (Placebo Comparator): Placebo administered IV every 2 weeks for a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8226 — MK-8226 administered IV at a weight-based dose every 2 weeks for 12 weeks.
  Arms: Part 1: MK-8226 0.3 mg/kg; Part 1: MK-8226 1 mg/kg; Part 1: MK-8226 10 mg/kg; Part 1: MK-8226 3 mg/kg; Part 2: MK-8226 3 mg/kg
Drug: Placebo — Placebo administered IV every 2 weeks for a period of 12 weeks.
  Arms: Part 1: Placebo (pooled); Part 2: Placebo

SUMMARY:
This is a 3-part study to assess the safety, tolerability, efficacy, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of MK-8226 in participants with moderate to severe atopic dermatitis. Part 1 (multiple rising dose study) objectives were to find the maximum tolerated dose (MTD) of MK-8226 and to assess safety and PK. Part 2 objectives were to determine safety, PK, and preliminary efficacy. Part 3 objectives were to further define safety and PK, and explore MK-8226 PK/PD to model the optimal dose range for future studies. The study was terminated early due to business reasons on 08 May 2014; final results from an analysis for Part 1 (efficacy, PK, safety, immunogenicity) and Part 2 (safety, immunogenicity) are summarized.

DETAILED DESCRIPTION:
Part 1 of the study is a multiple rising dose assessment of the safety, tolerability, and pharmacokinetics of MK-8226 for a period of 12 weeks followed by a 20-week off-treatment follow-up period.

Part 2 of the study is an assessment of the safety, tolerability, and efficacy of MK-8226 for 12 weeks followed by a 20-week off-treatment follow-up period.

In Part 3 of the study, participants will be treated with MK-8226 for a period of 12 weeks followed by a 20-week off-treatment follow-up period to evaluate pharmacokinetic and pharmacokinetic correlations to assist with modeling the dose range planned for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >=40 kg
* Clinical diagnosis of atopic dermatitis for at least 6 months prior
* Candidate for systemic or phototherapy (i.e., failed topical treatment)
* Moderate-to-severe disease as defined by Body Surface Area (BSA) ≥10%, EASI ≥12, and IGA ≥3
* No clinically significant abnormality on electrocardiogram
* No history of active or latent tuberculosis (TB) and no signs or symptoms suggestive of TB
* No history of active or latent TB and no signs or symptoms suggestive of TB
* History of inadequate response to a stable (≥ 1 month) regimen of topical corticosteroids or calcineurin inhibitors within 3 months before the screening visit

Exclusion Criteria:

* Concurrent significant skin disease
* Any significant organ dysfunction within 6 months prior
* History of clinically significant heart disease
* History of neoplastic disease
* Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Infection requiring oral antibiotics within 2 weeks prior
* Receipt of a live virus vaccine within 4 weeks prior
* Inability to refrain from topical or systemic therapy during course of the study
* Had major surgery or donated or lost >=1 unit of blood within 4 weeks prior
* Participation in another study within 4 weeks prior
* Current or regular user of illicit drugs or a history of drug or alcohol abuse within 1 year prior
* Pregnant, breast-feeding, or anticipated to conceive during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2014-10-20 (Actual); Study Completion 2014-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for study eligibility over 4 weeks prior to first dosing. Additional inclusion and exclusion criteria applied.
Period: Overall Study
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Started | 9 | 9 | 8 | 10 | 8 | 13 | 8
Completed | 8 | 4 | 4 | 5 | 3 | 0 | 0
Not Completed | 1 | 5 | 4 | 5 | 5 | 13 | 8
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1 | 5 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 1 | 0 | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo | Total
Number analyzed (Participants) | 9 | 9 | 8 | 10 | 8 | 13 | 8 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 8 | 10 | 8 | 13 | 8 | 64
  >=65 years | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (11.8) | 30.8 (13.4) | 41.6 (12.6) | 34.7 (10.2) | 37.8 (14.2) | 38.3 (11.5) | 33.9 (12.9) | 38.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 6 | 5 | 8 | 3 | 32
  Male | 5 | 7 | 4 | 4 | 3 | 5 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 32 Weeks
Population: The All Subjects as Treated (ASaT) population defined as all participants who received at least one dose of investigational drug was used for analysis.
Measure: Number; unit: participants
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 10 | 8 | 13 | 8
participants | 8 | 6 | 6 | 7 | 7 | 10 | 7

2. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to 12 Weeks
Population: The ASaT population defined as all participants who received at least one dose of investigational drug was used for analysis.
Measure: Number; unit: participants
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 10 | 8 | 13 | 8
participants | 0 | 1 | 1 | 0 | 0 | 0 | 1

3. Primary Outcome: Change From Baseline in the Eczema Area and Severity Index (EASI) for Study Part 1
Description: Reduction from baseline in EASI at Week 12 (interim analysis data). The EASI assesses intensity of four lesion characteristics (erythema, infiltration/population, excoriation, lichenification) each rated on a scale of 0 (absent) to 3 (severe) across four regions (head, trunk, upper and lower extremities). Affected areas in each region are assessed as percentage of body surface (head [10%], trunk [30%], upper extremities [20%], and lower extremities [40%]). The total score is a sum of each region score and can range from 0 (absent disease) to 72 (severe disease).
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) defined as all randomized subjects who received at least one dose of study treatment with baseline and at least one post-dose assessment (EASI) was used for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled)
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 5
Score on a scale | -5.77 (6.17) | -8.40 (9.39) | -10.20 (7.23) | -7.78 (8.35) | -0.38 (6.37)
Statistical Analysis 1: Comparison: Part 1: MK-8226 3 mg/kg vs Part 1: Placebo (Pooled); The reduction from baseline in EASI at week 12 for participants receiving MK-8226 3 mg/kg was compared to placebo (MK-8226 3 mg - Placebo). The constrained longitudinal data analysis model used variance component covariance matrix to model correlation among repeated visits, without adjustment for interaction of treatment group by visit; Test type: Superiority or Other; p = 0.015, Constrained longitudinal data analysis; Mean Difference (Final Values) = -9.82, 95% CI 2-sided [-16.87 to -2.77]

4. Secondary Outcome: Plasma Chemokine (C-C Motif) Ligand 17 (CCL17) Level in Study Part 2
Description: CCL17 is a pro-allergic chemokine that is assessed in human plasma. Levels of CCL17 are increased in allergic disease states.
Time Frame: Baseline, 48 Hours, Week 2, Week 4, Week 12, Week 16
Population: No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from Baseline [BL] in EASI) did not demonstrate adequate effect in an interim futility analysis. The study was early terminated from a business perspective.
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Plasma Chemokine (C-C Motif) Ligand 22 (CCL22) Level in Study Part 2
Description: CCL22 is a pro-allergic chemokine that is assessed in human plasma. Levels of CCL22 are increased in allergic disease states.
Time Frame: Baseline, 48 Hours, Week 2, Week 4, Week 12, Week 16
Population: No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis. The study was early terminated from a business perspective.
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Area Under the Concentration-time Curve of MK-8226 From Time 0 to Tau (AUC0-tau) Following Multiple Intravenous Dose Administration
Description: AUC(0-tau) defined as AUC from time zero to tau where tau is the dosing interval (312 hours) was determined for the first and last periods of MK-8226 dosing. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 1 (incl. predose), 3, 5, 9, 14 (incl. predose), 70 (incl. predose), 72, 74, 84. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 1, 3, 5, 9, 14, 70, 72, 74, 84
Population: The Per-Protocol (PP) population defined as all participants compliant with study procedure with data available (AUC0-tau) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 9 | 7 | 8 | 10
μg*hr/mL
  Week 1 (n=9,7,8,10) | 1000 (18.2) | 3300 (29.3) | 9300 (19.1) | 31400 (11.2)
  Week 10 (n=8,5,6,6) | 2310 (11) | 8530 (15.4) | 21100 (28.8) | 82100 (16.2)

7. Secondary Outcome: AUC From Time 0 to Last Measurement (AUC0-last) of MK-8226 Following Multiple Intravenous Dose Administration
Description: AUC0-last defined as AUC up to the last measured concentration was determined for the last period of dosing (starting Week 10 [Day 70]) up to the last measurement. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 70 (incl. predose), 72, 74, 84, 98, 112, 140, 168, 196, and 224. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 70, 72, 74, 84, 98, 112, 140, 168, 196, 224
Population: The PP population defined as all participants compliant with study procedure with data available (AUC0-last) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 8 | 6 | 6 | 6
μg*hr/mL | 6460 (34.3) | 22600 (65.8) | 47100 (97.2) | 264000 (25.2)

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of MK-8226 Following Multiple Dose Intravenous Administration
Description: Cmax was determined for the first and last periods of MK-8226 dosing. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 1 (incl. predose), 3, 5, 9, 14 (incl. predose), 70 (incl. predose), 72, 74, and 84. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 1, 3, 5, 9, 14, 70, 72, 74, 84
Population: The PP population defined as all participants compliant with study procedure with data available (Cmax) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 9 | 8 | 8 | 10
μg/mL
  Week 1 (n=9,8,8,10) | 7.12 (21.9) | 21.6 (26.0) | 60.3 (18.0) | 200 (12.1)
  Week 10 (n=8,6,6,6) | 11.7 (9.63) | 42.4 (20.1) | 106 (19.6) | 398 (17.1)

9. Secondary Outcome: Clearance (CL) of MK-8226 Following Multiple Dose Intravenous Administration
Description: CL, the volume of plasma cleared of drug per unit time, was determined for the last period of dosing (starting Week 10 [Day 70]) in the treatment period. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 1 (incl. predose), 3, 5, 9, 14 (incl. predose), 28 (incl. predose), 42 (incl. predose), 56 (incl. predose), 70 (incl. predose), 72, 74, and 84. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 1, 3, 5, 9, 14, 28, 42, 56, 70, 72, 74, 84
Population: The PP population defined as all participants compliant with study procedure with data available (CL) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day/kg
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 8 | 5 | 6 | 6
mL/day/kg | 3.04 (11) | 2.81 (15.4) | 3.33 (28.8) | 2.9 (16.2)

10. Secondary Outcome: Volume of Distribution (Vd) of MK-8226 Following Multiple Intravenous Administration
Description: Vd, a theoretical approximation of degree to which the drug distributes in body tissue rather than plasma (higher Vd indicates greater tissue distribution), was determined for the last period of dosing (starting Week 10 [Day 70]) in the treatment period. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 70 (incl. predose), 72, 74, 84, 98, 112, 140, 168, 196, and 224. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 70, 72, 74, 84, 98, 112, 140, 168, 196, 224
Population: The PP population defined as all participants compliant with study procedure with data available (Vd) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 8 | 5 | 4 | 6
mL/kg | 103 (27.6) | 122 (26.8) | 102 (62.1) | 120 (25.3)

11. Secondary Outcome: Terminal Half Life (t1/2) of MK-8226 Following Multiple Dose Intravenous Administration
Description: t1/2, the time needed for the concentration of drug to reach half the initial concentration, was determined for the last period of dosing (starting Week 10 [Day 70]) up to the last measurement. MK-8226 was administered on Days 1, 14, 28, 42, 56, and 70. Blood concentrations of MK-8226 were determined on Days 70 (incl. predose), 72, 74, 84, 98, 112, 140, 168, 196, and 224. The placebo group is not included; this endpoint evaluated only the MK-8226 groups. No analysis was performed for Part 2 non-safety secondary endpoints after the Part 1 primary endpoint (Change from BL in EASI) did not demonstrate adequate effect in an interim futility analysis.
Time Frame: Days 70, 72, 74, 84, 98, 112, 140, 168, 196, 224
Population: The PP population defined as all participants compliant with study procedure with data available (t1/2) from at least one treatment was used for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg
Number analyzed (Participants) | 8 | 5 | 4 | 6
days | 23.6 (33.5) | 30 (15.9) | 24.7 (51.3) | 28.7 (15.7)

12. Secondary Outcome: Change From Baseline in the Eczema Area and Severity Index (EASI) for Study Part 2
Description: The EASI assesses intensity of four lesion characteristics (erythema, infiltration/population, excoriation, lichenification) each rated on a scale of 0 (absent) to 3 (severe) across four regions (head, trunk, upper and lower extremities). Affected areas in each region are assessed as percentage of body surface (head [10%], trunk [30%], upper extremities [20%], and lower extremities [40%]). The total score is a sum of each region score and can range from 0 (absent disease) to 72 (severe disease).
Time Frame: Baseline, Week 4, Week 8, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of Clear or Almost Clear in Study Part 2
Description: Percentage of participants achieving an IGA of atopic dermatitis of "clear-0" or "almost clear-1". The IGA is a six-point scale measuring the severity of disease at time of physical examination of the participant by the physician. The IGA is scored 0 (Clear) to 5 (Very severe disease).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the Scoring Atopic Dermatitis Scale (SCORAD) in Study Part 2
Description: The SCORAD index scale combines 1) intensity of six lesion characteristics (erythema, edema/papulation, oozing/crusts, excoriations, lichenification, dryness) as assessed by the physician on a scale of 0 (absent) to 3 (severe) across four regions (head, trunk, upper and lower extremities) along with 2) subjective symptoms of pruritus and sleep disturbance as reported by the patient on a visual analog scale (VAS) from 1 to 10 cm (increasing severity). Physician assessment of affected areas in each region is made as percentage of body surface (head [10%], trunk [30%], upper extremities [20%], and lower extremities [40%]). The final SCORAD index score, ranging from 0 (absent disease) to 103 (severe disease), is calculated according to the weighted formula: (0.2 x area) + (3.5 x [sum of intensity score for each of the 6 items]) + participant's subjective score.
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline in Participant Pruritus in Study Part 2
Description: Skin pruritus (itching) is a typical characteristic of atopic dermatitis. Participant subjective assessment of pruritus (component of SCORAD) is rated on a VAS ranging from 1 to 10 cm (increasing severity).
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Participant Sleep Disturbance in Study Part 2
Description: Sleep disturbance (sleep loss, disruption, or interference) due to unremitting pruritus and other causes is a quality of life issue in moderate to severe atopic dermatitis. Participant subjective assessment of sleep disturbance (component of SCORAD) over the past 3 days is rated on a VAS ranging from 1 to 10 cm (increasing severity).
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants Requiring As-Needed Oral Antihistamines as Rescue Medication in Study Part 2
Description: Oral antihistamines (i.e., diphenhydramine, acrivastine fenistil) were provided as as-needed rescue medication for severe pruritus.
Time Frame: Up to Week 12
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Change From Baseline in the Participant's Global Impression of Disease Status in Study Part 2
Description: Participant subjective impression of improvement of his/her disease condition is scored on a six-point scale: 0 (Clear) to 5 (Very severe disease).
Time Frame: Baseline, Week 4, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Percentage of Participants With >=50% Improvement in EASI Score
Description: as for outcome 12
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 5
Arm/Group | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibody (ADA) Formation
Description: Testing for ADA positivity and neutralizing response and antibody titre quantification are performed with blood (serum) samples collected at baseline (Day 1 predose) and Days 14, 28, 42, 56, 74, 112, and 224. Neutralizing response refers to ADA neutralizing interference with study drug assessed in vitro. Non-Treatment emergent ADA refers to presence of ADAs (as determined by assay) in the absence of treatment with study drug (i.e., at predose).
Time Frame: Days 1 (predose) and Days 14, 28, 42, 56, 74, 112, and 224
Population: The ADA evaluable population defined as all participants with at least one ADA sample available after treatment with MK-8226 or placebo was used for analysis.
Measure: Number; unit: Participants
Groups:
- Part 1: Placebo (Pooled): Dose-matched placebo administered IV every 2 weeks for a period of 12 weeks. No participant met criteria for inclusion in the evaluable population.
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 0 | 12 | 2
Participants
  Non Treatment emergent ADA positive | 0 | 1 | 0 | 0 |  | 0 | 0
  Treatment emergent ADA positive | 0 | 0 | 1 | 0 |  | 2 | 0
  ADA positive: Max titer 1:10 | 0 | 0 | 0 | 0 |  | 0 | 0
  ADA positive: Max titer 1:50 | 0 | 0 | 1 | 0 |  | 1 | 0
  ADA positive: Neutralizing response positive | 0 | 0 | 1 | 0 |  | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 32 Weeks
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Groups:
- Part 1: MK-8226 0.3 mg/kg; Part 1: MK-8226 1 mg/kg; Part 1: MK-8226 3 mg/kg; Part 1: MK-8226 10 mg/kg; Part 2: MK-8226 3 mg/kg: MK-8226 administered IV at a weight-based dose every 2 weeks for a period of 12 weeks.
Arm/Group | Part 1: MK-8226 0.3 mg/kg | Part 1: MK-8226 1 mg/kg | Part 1: MK-8226 3 mg/kg | Part 1: MK-8226 10 mg/kg | Part 1: Placebo (Pooled) | Part 2: MK-8226 3 mg/kg | Part 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 1/10 | 0/8 | 0/13 | 1/8
Other Adverse Events (participants affected / at risk) | 8/9 | 6/9 | 6/8 | 7/10 | 7/8 | 10/13 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-8226 0.3 mg/kg (N=9) | Part 1: MK-8226 1 mg/kg (N=9) | Part 1: MK-8226 3 mg/kg (N=8) | Part 1: MK-8226 10 mg/kg (N=10) | Part 1: Placebo (Pooled) (N=8) | Part 2: MK-8226 3 mg/kg (N=13) | Part 2: Placebo (N=8)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-8226 0.3 mg/kg (N=9) | Part 1: MK-8226 1 mg/kg (N=9) | Part 1: MK-8226 3 mg/kg (N=8) | Part 1: MK-8226 10 mg/kg (N=10) | Part 1: Placebo (Pooled) (N=8) | Part 2: MK-8226 3 mg/kg (N=13) | Part 2: Placebo (N=8)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palatal swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gravitational oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 4 (5) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 1 (2) | 3 (4) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.